CLINICAL TRIAL: NCT00788723
Title: Cortical Excitability in Patients With Severe Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Natallia Lapitskaya, MD, Hammel Neurorehabilitation and Research Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HNRC-AAU-08-1
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2008-11

CONDITIONS: Severe Traumatic Brain Injury; Subarachnoid Hemorrhage; Anoxic Brain Injury
Keywords: Severe Brain Injury; Excitability; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Hypoxia-Ischemia, Brain; Brain Injuries | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Patients with severe brain injury, awake, but have cognitive problems
  Interventions: Device: Transcranial Magnetic Stimulation
- 2 (Experimental): Patients with severe brain injury and disorders of consciousness ( in minimally conscious or in vegetative state)
  Interventions: Device: Transcranial Magnetic Stimulation
- 3 (Experimental): Healthy volunteers
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial magnetic stimulation (TMS) using paired-pulse technique at different interstimulus intervals (ISIs) allows the study of the excitatory and inhibitory system of human motor cortex non-invasively. Motor evoked potentials (MEP) will be recorded, and stored on a VikingSelect (Viasys Healthcare, USA). Two magnetic stimulators (Magstim 200, The Magstim Company Ltd, U.K.) connected through a Bistim and a Magstim figure-of-eight coil will be used for TMS.
  Other Names: Paired-pulse transcanial magnetic stimulation

SUMMARY:
The aim of the study is to evaluate the cortical excitability in the severe brain injured patients. We hypothesize that:

1. There is a continuous decrease in intracortical inhibition from healthy subjects to awake patients with severe brain injury, and to patients with impaired consciousness.
2. Decreased intracortical inhibition correlate with the degree of impairment assessed with the clinical scores in patients with severe brain injury.

DETAILED DESCRIPTION:
Design: Prospective controlled non-randomized study. Materials and methods: 30 patients with severe brain injury and 15 healthy volunteers will be included in this study.

The study design is illustrated below:

1. Clinical assessment (Rancho Los Amigos Scale, Functional Independence Measure, Early Functional Abilities).
2. Somatosensory Evoked Potentials.
3. Transcranial Magnetic Stimulation: single and paired stimulation protocols.

Statistical evaluation: All collected data will be tested with reference to normal distribution. If the data is not distributed normally, then we will use either a logarithmic transformation before we use parametric statistics, or we will use non-parametric statistics for further calculations.Further analysis of the data will be done with the help of variance analysis with an inter-individually factor as a group (awake patients vs patients with disorders of consciousness vs control persons) and intra-individually factors as 1) interstimulus intervals for transcranial magnetic stimulation and clinical scores (RLAS vs FIM vs EFA).

Significance level is set to 0.05 for all effect parameters.

ELIGIBILITY:
Inclusion Criteria:

1. severe brain injury (Glasgow Coma Scale score (GCS) less than 8 on admission to the acute hospital);
2. stable vital functions;
3. age over 18 years old;
4. informed content from patient/relatives/legal guardian.

Exclusion Criteria:

1. other neurological diseases than brain injury;
2. pregnancy;
3. TMS contraindications (epilepsy, metallic implantants: pacemaker or medicine pump, ferromagnetic or electronically operated stapedial implants, haemostatic clips, metallic splinters in the orbit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-03 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Short Afferent Inhibition | Within one week after clinical assessment

SECONDARY OUTCOMES:
Short Intracortical Inhibition | Within one week after clinical assessment
Intracortical Facilitation | Within one week after clinical assessment
Motor threshold | Within one week after clinical assessment

CONTACTS AND LOCATIONS:
Overall Officials: Natallia Lapitskaya, MD, Principal Investigator — Hammel Neurorehabilitation and Research Centre
Locations (1):
- Hammel Neurorehabilitation and Research Centre, Hammel, Denmark